CLINICAL TRIAL: NCT03669120
Title: Tailored or Non-Tailored Smoking Cessation Intervention for Sexual and Gender Minorities
Brief Title: Tailored Smoking Cessation Intervention in Promoting Sexual and Gender Minority Smokers to Quit Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0564; NCI-2018-01821 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0564 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Cigarette Smoker; Current Every Day Smoker

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (mainstream instructional care) (Active Comparator): Participants receive mainstream instructional care including brief advice on how to quit smoking, 10-week supply of NRT in the form of nicotine patches, and intensive print materials to promote smoking cessation.
  Interventions: Other: Informational Intervention
- Arm II (tailored intensive care) (Experimental): Participants receive tailored intensive care including brief advice on how to quit smoking, NRT, and intensive print materials to promote smoking cessation as in Arm I. Participants also receive individualized text based messages to promote smoking cessation for 6 months.
  Interventions: Other: Informational Intervention; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Other: Informational Intervention — Receive advice to quit smoking and materials to promote smoking cessation
Behavioral: Telephone-Based Intervention — Receive individualized text based messages
  Arms: Arm II (tailored intensive care)

SUMMARY:
This trial studies how well tailored smoking cessation intervention works in promoting sexual and gender minority smokers to quit smoking. A program that is specifically designed for the lesbian, gay, bisexual, and transgender community may affect these participants differently than a traditional approach.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the feasibility of two different approaches for smoking cessation (print materials developed for smoking cessation among the mainstream population versus [vs.] an individualized text based approach) among 60 lesbian, gay, bisexual, and transgender (LGBT) smokers.

SECONDARY OBJECTIVES:

I. To assess the levels of helpfulness, appropriateness, and perceived difficulty of the above mentioned cessation approaches among 60 LGBT smokers.

EXPLORATORY OBJECTIVES:

I. To test the smoking abstinence rates of two different individualized intensive cessation approaches (mainstream vs. individually-tailored) among 60 LGBT smokers.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive mainstream instructional care including brief advice on how to quit smoking, 10-week supply of nicotine replacement therapy (NRT) in the form of nicotine patches, and intensive print materials to promote smoking cessation.

ARM II: Participants receive tailored intensive care including brief advice on how to quit smoking, NRT, and intensive print materials to promote smoking cessation as in Arm I. Participants also receive individualized text based messages to promote smoking cessation for 6 months.

After completion of study, participants are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female owning a cell phone with a reachable contact number
* Self-identified as LGBT individual, regardless human immunodeficiency virus (HIV) serologic status
* Smoked at least 100 cigarettes in lifetime
* Currently smoking at least 5 cigarettes a day, on average
* Willing to set a quit smoking date within a week of the enrollment
* English speaking

Exclusion Criteria:

* Expired carbon monoxide (CO) levels below 7 ppm
* Positive history of a medical condition that precludes use of the nicotine patch (e.g., recent myocardial infarction, significant skin disorder, previous severe adverse reaction to nicotine patch, pregnant or breast feeding, assessed with our standard protocol for determining NRT eligibility)
* Current use of NRT or other smoking cessation medications (e.g., varenicline or bupropion)
* Pregnant or nursing
* Enrolled in another smoking cessation program
* Partner enrolled on current study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Computing recruitment rate | At baseline
  Will be summarized using descriptive statistics such as the mean, standard deviation, median, interquartile range, and frequency where appropriate. Confidence intervals of 90% for the participating rates at baseline and retention rates at 3- and 6- follow-up will be provided.
Retention rates | At 3 and 6 months
  Will be summarized using descriptive statistics such as the mean, standard deviation, median, interquartile range, and frequency where appropriate. Confidence intervals of 90% for the participating rates at baseline and retention rates at 3- and 6- follow-up will be provided.

SECONDARY OUTCOMES:
Levels of helpfulness | Up to 6 months
  Will be measured by asking: "Were the text messages helpful in your attempt to quit smoking cigarettes?" (Likert scale from 0= Not at all helpful to 4=Very helpful). Will use t-test to compare between arms.
Appropriateness | Up to 6 months
  Will be measured by asking: "Regarding the number of text messages received per day, did you think that there were:" (Likert scale from 0=Too many to 2=Not enough). Will use t-test to compare between arms.
Perceived difficulty | Up to 6 months
  Will be measured by asking: "How easy was it to view the text messages?" (Likert scale from 0=Not at all easy to 4=Very easy) "How easy was it to respond to the text messages?" (Likert scale from 0=Not at all easy to 4=Very easy). Will use t-test to compare between arms.

OTHER OUTCOMES:
Point prevalence abstinence | Up to 6 months
  Seven day smoking abstinence along with negative saliva cotinine will be the primary definition of smoking abstinence for this study. Important covariates that will be used to adjust for potential baseline differences include level of education, biological sex, marital status, gender identity, race, working status, income, years smoking, smoking initiation, use of other tobacco products, and living with other household members who smoke.
Salivary cotinine assessed by NicAlert test | Up to 6 months
  Important covariates that will be used to adjust for potential baseline differences include level of education, biological sex, marital status, gender identity, race, working status, income, years smoking, smoking initiation, use of other tobacco products, and living with other household members who smoke.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Tami-Maury, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org